CLINICAL TRIAL: NCT00737048
Title: A Double-Blind Comparative Study of JNS013 in Patients With Post-Tooth-Extraction Pain
Brief Title: A Comparative Study of JNS013 in Participants With Post-Tooth-Extraction Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR015109; JNS013-JPN-03
Record Dates: First submitted 2008-08-14; First posted 2008-08-18 (Estimated); Results first posted 2013-08-01 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Pain; Postoperative Pain
Keywords: Pain; Tooth extraction; Oral surgery; Postoperative pain; JNS013; Tramadol hydrochloride; Acetaminophen
MeSH Terms: conditions — Pain; Pain, Postoperative | interventions — Tramadol; Acetaminophen

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tramadol plus Acetaminophen and Placebo (Experimental): Tramadol hydrochloride and acetaminophen combination tablet will be administered as single oral dosing of two tablets at a dose of 75 and 650 milligram respectively, along with two oral capsules of matching placebo, within 30 minutes after the intensity of pain associated with tooth extraction showed greater than or equal to (>=) 50.0 millimeter (mm) on the Visual Analog Scale (VAS), score ranging from 0 mm (no pain) to 100 mm (worst possible pain).
  Interventions: Drug: Placebo; Drug: Tramadol plus Acetaminophen
- Tramadol and Placebo (Experimental): Tramadol hydrochloride will be administered as single oral dosing of two capsules once at a dose of 75 milligram, along with two oral tablets of matching placebo, within 30 minutes after the intensity of pain associated with tooth extraction showed >= 50.0 mm on the VAS, score ranging from 0 mm (no pain) to 100 mm (worst possible pain).
  Interventions: Drug: Tramadol Hydrochloride; Drug: Placebo
- Acetaminophen and Placebo (Experimental): Acetaminophen will be administered as single oral dosing of two capsules once at a dose of 650 milligram, along with two oral tablets of matching placebo, within 30 minutes after the intensity of pain associated with tooth extraction showed >= 50.0 mm on the VAS, score ranging from 0 mm (no pain) to 100 mm (worst possible pain).
  Interventions: Drug: Acetaminophen; Drug: Placebo

INTERVENTIONS:
Drug: Tramadol Hydrochloride — Tramadol hydrochloride two oral capsules will be administered once as 75 milligram (mg).
  Arms: Tramadol and Placebo
Drug: Acetaminophen — Acetaminophen two oral capsules will be administered once as 650 mg.
  Arms: Acetaminophen and Placebo
Drug: Placebo — Two oral tablets or capsules of matching Placebo will be administered once along with Tramadol Hydrochloride and/or acetaminophen.
Drug: Tramadol plus Acetaminophen — Tramadol hydrochloride and acetaminophen combination tablet will be administered as single oral dosing of two tablets at a dose of 75 and 650 milligram respectively.
  Other Names: JNS013
  Arms: Tramadol plus Acetaminophen and Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of JNS013 with single oral dose administration in participants with pain after tooth-extraction of mandibular impacted wisdom tooth.

DETAILED DESCRIPTION:
This is a multi-center (conducted in more than one center), double-blind (neither Physician nor participant knows the name of the assigned drug), randomized (study drug assigned by chance), parallel-group (each group of participant will be treated at the same time) and comparative study in participants having pain intensity of at least 50.0 millimeter (mm) (on visual analog scale, score ranging from 0 mm [no pain] to 100 mm [worst possible pain]), following extraction of an impacted mandibular wisdom tooth. The study consists of 3 parts: Pre-observation (7 days before study commences on Day 1); Treatment (Day 1, consists of single oral dosing of either tramadol plus acetaminophen and placebo; or tramadol and placebo; or acetaminophen and placebo) and Follow-up (Day 2 and 8). All the eligible participants will be randomly assigned to 1 of the 3 study treatments. Efficacy of the participants will primarily be evaluated through total pain relief, which will be evaluated on numerical rating scale. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants planned to receive a tooth extraction of one mandibular impacted wisdom tooth
* Participants who require bone removal and separation of the crown at tooth extraction
* Participants whose intensity of pain associated with tooth extraction within 2 hours after tooth extraction is greater than or equal to 50.0 millimeter on the visual analog scale (VAS)
* Participants who did not undergo general anesthesia or sedation at tooth extraction
* Participants without an abnormality (including laboratory test values) corresponding to Grade 3 in the "Criteria for severity classification of adverse drug reactions" during the pretreatment observation period

Exclusion Criteria:

* Participants with conditions for which tramadol is contraindicated
* Participants with conditions for which acetaminophen is contraindicated
* Participants with history of convulsions or the possibility of convulsive seizures
* Pregnant participants or those who may be pregnant, lactating mothers, and those who wish pregnancy during the study period
* Participants with concurrent, previous, or possible alcohol dependence, drug dependence or narcotic addiction

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 328 (Actual)
Dates: Start 2008-03; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K., Japan Clinical Trial, Study Director — Janssen Pharmaceutical K.K.
Locations (11):
- Japan (11):
  - Isehara
  - Kitakyushu
  - Kumamoto
  - Ohta-Ku
  - Osaka
  - Sapporo
  - Shimotsuga
  - Shimotsuke
  - Tokyo
  - Yokohama
  - Yokosuka

REFERENCES:
- See also: A confirmatory study of JNS013 in patients with post-tooth-extraction pain — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=422&filename=CR015109_CSR.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Tramadol Hydrochloride Plus Acetaminophen and Placebo: Tramadol hydrochloride and acetaminophen combination tablet was administered as 75 and 650 milligram respectively, as single oral dose of two tablets, along with two oral capsules of matching placebo, within 30 minutes after the intensity of pain associated with tooth extraction showed greater than or equal to (>=) 50.0 millimeter (mm) on the Visual Analog Scale (VAS), score ranging from 0 mm (no pain) to 100 mm (worst possible pain).
- Tramadol Hydrochloride and Placebo: Tramadol hydrochloride was administered as 75 milligram, as single oral dose of two capsules, along with two oral tablets of matching placebo, within 30 minutes after the intensity of pain associated with tooth extraction showed >= 50.0 mm on the VAS, score ranging from 0 mm (no pain) to 100 mm (worst possible pain).
- Acetaminophen and Placebo: Acetaminophen was administered as 650 milligram as single oral dose of two capsules, along with two oral tablets of matching placebo, within 30 minutes after the intensity of pain associated with tooth extraction showed >= 50.0 mm on the VAS, score ranging from 0 mm (no pain) to 100 mm (worst possible pain).
Period: Overall Study
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Started | 132 | 66 | 130
Completed | 129 | 60 | 126
Not Completed | 3 | 6 | 4
Not completed — Physician Decision | 0 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0
Not completed — Worsening of the symptoms | 3 | 5 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo | Total
Number analyzed (Participants) | 132 | 66 | 130 | 328
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.1 (8.3) | 27.8 (8.6) | 27.5 (8.2) | 27.8 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 61 | 32 | 66 | 159
  Male | 71 | 34 | 64 | 169
Visual Analog Scale (VAS) Score [Mean (Standard Deviation); unit: Units on a scale] — Pain was assessed by using Visual Analogue Scale (VAS) score ranges from 0 millimeter (mm)=no pain to 100 mm=worst possible pain. An increase in score from Baseline represented disease progression and decrease represented treatment response.
  Units on a scale | 62.28 (9.85) | 60.33 (7.63) | 61.32 (8.81) | 61.51 (9.04)

OUTCOME MEASURES:

1. Primary Outcome: Total Pain Relief Based on Numerical Rating Scale (NRS) Score
Description: Total pain relief was evaluated using numerical rating scale score ranging from 0 to 32, wherein 0 indicates no treatment response and 32 indicates the most improved. Higher score indicates treatment response.
Time Frame: 8 hours
Population: Final analysis set (FAS) population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale | 17.7 (7.91) | 12.4 (8.36) | 13.3 (8.07)
Statistical Analysis 1: Comparison: Tramadol Hydrochloride Plus Acetaminophen and Placebo vs Tramadol Hydrochloride and Placebo; Statistical Analysis 1 for Total pain relief based on numerical rating scale score; Test type: Superiority or Other; p < 0.0001, Fisher Least Signiﬁcant Diﬀerence Method; Mean Difference (Final Values) = -5.3, Standard Deviation 8.06
Statistical Analysis 2: Comparison: Tramadol Hydrochloride Plus Acetaminophen and Placebo vs Acetaminophen and Placebo; Statistical Analysis 2 for Total pain relief based on numerical rating scale score; Test type: Superiority or Other; p < 0.0001, Fisher Least Signiﬁcant Diﬀerence Method; Mean Difference (Final Values) = -4.3, Standard Deviation 7.99

2. Secondary Outcome: Total Pain Relief Based on Numerical Rating Scale (NRS) Score Every 4 Hours up to 8 Hours
Description: as for outcome 1
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale
  0-4 hours | 9.6 (3.90) | 6.3 (4.11) | 7.4 (3.97)
  4-8 hours | 8.0 (4.73) | 6.1 (4.67) | 5.9 (4.71)

3. Secondary Outcome: Sum of Pain Intensity Difference (SPID)
Description: Pain Intensity (PI) was assessed using numerical rating scale score ranging from 0 to 32, wherein 0 indicates no treatment response and 32 indicates the most improved. Scores were measured at Baseline (that is, 0 hours after tooth extraction) and 8 hours post-administration of study treatments.Pain intensity difference (PID) was calculated (that is, for 0-8 hours, time point [8 hour] score minus baseline [0 hour] score).
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale | 6.4 (5.90) | 2.9 (5.12) | 4.1 (5.84)

4. Secondary Outcome: Sum of Pain Relief Combined With Pain Intensity Difference (SPRID)
Description: The SPRID is the sum of pain relief scores combined with pain intensity difference, score ranging from from (-) 24 (the worst) through 56 (the most improved). Higher score indicates treatment response. Pain Intensity (PI) and Pain relief (PAR) were assessed using numerical rating scale score ranging from 0 to 32, wherein 0 indicates no treatment response and 32 indicates the most improved. Scores were measured at Baseline (that is, 0 hours after tooth extraction) and at 8 hours post-administration of study treatments. Pain intensity difference (PID) was calculated (that is, for 0-8 hours, time point [8 hour] score minus baseline [0 hour] score).
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale | 24.0 (13.03) | 15.3 (12.43) | 17.4 (13.17)

5. Secondary Outcome: Change From Baseline in Visual Analog Scale (VAS) Score at 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 Hours Post-administration of Study Treatment
Description: Pain was assessed by using Visual Analogue Scale (VAS) score ranges from 0 millimeter (mm)=no pain to 100 mm=worst possible pain. An increase in score from Baseline represented disease progression and decrease represented treatment response.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale
  Change at Hour 0.5 | -22.11 (23.466) | -4.28 (20.001) | -15.50 (22.336)
  Change at Hour 1 | -36.79 (23.603) | -12.82 (27.372) | -26.68 (24.570)
  Change at Hour 2 | -42.71 (23.631) | -20.94 (27.904) | -28.43 (27.583)
  Change at Hour 3 | -41.40 (26.707) | -25.75 (28.509) | -28.40 (30.544)
  Change at Hour 4 | -37.70 (27.266) | -21.75 (29.870) | -24.83 (30.753)
  Change at Hour 5 | -34.78 (28.173) | -17.56 (29.110) | -21.48 (31.350)
  Change at Hour 6 | -30.20 (30.932) | -15.70 (31.033) | -17.51 (31.875)
  Change at Hour 7 | -26.37 (32.456) | -13.18 (30.335) | -15.62 (32.562)
  Change at Hour 8 | -22.85 (33.116) | -13.03 (30.916) | -14.48 (32.638)

6. Secondary Outcome: Mean Change Over Time for Pain Intensity Difference (PID) at 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 Hours Post-Administration of Study Treatment
Description: The PID is defined as difference between current pain intensity (PI) and Baseline PI, PI was assessed using numerical rating scale score ranging from 0 to 32, wherein 0 indicates no treatment response and 32 indicates the most improved. Higher score indicates treatment response. Mean change from Baseline (that is, 0 hours after tooth extraction) at specified end time points were evaluated.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale
  PID:Change at Hour 0.5 | 0.6 (0.67) | 0.1 (0.55) | 0.5 (0.73)
  PID:Change at Hour 1 | 0.9 (0.71) | 0.4 (0.70) | 0.7 (0.72)
  PID:Change at Hour 2 | 1.1 (0.78) | 0.5 (0.71) | 0.8 (0.79)
  PID:Change at Hour 3 | 1.1 (0.87) | 0.5 (0.73) | 0.7 (0.84)
  PID:Change at Hour 4 | 0.9 (0.85) | 0.4 (0.70) | 0.6 (0.84)
  PID:Change at Hour 5 | 0.8 (0.85) | 0.3 (0.73) | 0.5 (0.88)
  PID:Change at Hour 6 | 0.7 (0.88) | 0.4 (0.80) | 0.4 (0.88)
  PID:Change at Hour 7 | 0.6 (0.92) | 0.2 (0.77) | 0.3 (0.93)
  PID:Change at Hour 8 | 0.5 (0.94) | 0.2 (0.77) | 0.3 (0.91)

7. Secondary Outcome: Mean Change Over Time for Pain Relief (PAR) at 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 Hours Post-administration of Study Treatment
Description: Pain Relief (PAR) was assessed using numerical rating scale score ranging from 0 to 32, wherein 0 indicates no treatment response and 32 indicates the most improved. Higher score indicates treatment response. Mean change from Baseline (that is, 0 hours after tooth extraction) at specified end time points were evaluated.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale
  PAR:Change at Hour 0.5 | 1.5 (1.12) | 0.7 (0.86) | 1.3 (0.99)
  PAR:Change at Hour 1 | 2.3 (1.08) | 1.4 (1.13) | 2.0 (1.11)
  PAR:Change at Hour 2 | 2.7 (1.06) | 1.7 (1.23) | 2.0 (1.18)
  PAR:Change at Hour 3 | 2.6 (1.18) | 1.9 (1.20) | 2.0 (1.21)
  PAR:Change at Hour 4 | 2.4 (1.22) | 1.7 (1.18) | 1.8 (1.20)
  PAR:Change at Hour 5 | 2.2 (1.21) | 1.6 (1.16) | 1.6 (1.27)
  PAR:Change at Hour 6 | 2.1 (1.20) | 1.6 (1.28) | 1.5 (1.25)
  PAR:Change at Hour 7 | 1.9 (1.30) | 1.5 (1.19) | 1.4 (1.27)
  PAR:Change at Hour 8 | 1.8 (1.30) | 1.5 (1.15) | 1.4 (1.25)

8. Secondary Outcome: Mean Change Over Time for Pain Relief Combined With Pain Intensity Difference (PRID) at 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 Hours Post-administration of Study Treatment
Description: Pain Relief combined with pain Intensity Difference (PRID) represented pain relief scores combined with Pain Intensity difference (PID) scores. PRID score ranges from -3 (the worst) through +7 (the most improved). Higher score indicates treatment response. Mean change from Baseline (that is, 0 hours after tooth extraction) at specified end time points were evaluated.
Time Frame: 0.5, 1, 2, 3, 4, 5, 6, 7 and 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Units on a scale
  PRID:Change at Hour 0.5 | 2.1 (1.67) | 0.8 (1.29) | 1.8 (1.61)
  PRID:Change at Hour 1 | 3.2 (1.68) | 1.8 (1.71) | 2.7 (1.69)
  PRID:Change at Hour 2 | 3.8 (1.71) | 2.2 (1.80) | 2.8 (1.85)
  PRID:Change at Hour 3 | 3.7 (1.92) | 2.4 (1.75) | 2.7 (1.92)
  PRID:Change at Hour 4 | 3.3 (1.95) | 2.1 (1.71) | 2.4 (1.92)
  PRID:Change at Hour 5 | 3.0 (1.93) | 1.9 (1.74) | 2.1 (2.03)
  PRID:Change at Hour 6 | 2.8 (1.96) | 1.9 (1.92) | 1.8 (2.00)
  PRID:Change at Hour 7 | 2.5 (2.12) | 1.7 (1.81) | 1.8 (2.08)
  PRID:Change at Hour 8 | 2.3 (2.12) | 1.7 (1.78) | 1.6 (2.04)

9. Secondary Outcome: Time to Reach the Onset of Drug Efficacy and Time to Recurrence of Pain After the Onset of Drug Efficacy
Description: Time to reach the onset of drug efficacy (TOE) means time took by participants for the onset of relief from pain after tooth-extraction and time to recurrence of pain (TOR) after the onset of drug efficacy (that is, duration of drug efficacy) were assessed after study drug treatment.
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data. 'N' (number of participants analyzed) signifies those participants who were evaluable for this measure & 'n' signifies those participants who were evaluable for this measure at given time points.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 102 | 36 | 104
Minutes
  TOE (n=102, 36, 104) | 47.6 (40.88) | 82.8 (82.88) | 53.5 (47.97)
  TOR (n=41, 14, 53) | 252.5 (119.03) | 207.9 (126.44) | 198.2 (120.24)

10. Secondary Outcome: Percentage of Participants With Categorical Score for Patient Impressions
Description: Percentage of participants with patient impressions were assessed on categories, that are: worked well; worked; worked a little; and didn't work.
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Number; unit: Percentage of participants
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Percentage of participants
  Worked well | 28.7 (10) | 16.4 (12.43) | 15.7 (13.17)
  Worked | 55.8 (6.29) | 44.3 (6.04) | 53.5 (6.39)
  Worked a little | 13.2 (7.73) | 24.6 (7.04) | 22.8 (7.69)
  Didn't work | 2.3 | 14.8 | 7.9

11. Secondary Outcome: Number of Participants Treated With a Relief Analgesic
Description: Participants who were treated with a relief analgesic were assessed. Analgesics are the compounds capable of relieving pain without the loss of consciousness.
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: FAS population included all the participants who received the study treatment and had efficacy assessment data.
Measure: Number; unit: Participants
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 132 | 66 | 130
Participants | 37 | 25 | 54

12. Secondary Outcome: Percentage of Participants With Treatment Response Based on Evaluation Criteria for Efficacy of Analgesics in Post-Tooth-Extraction Pain
Description: Percentage of participants were assessed with treatment response based on "evaluation criteria for efficacy of analgesics in post-tooth-extraction pain" for the efficacy of analgesics used to treat pain following tooth extraction. Participants were assessed as "very effective, effective, somewhat effective and ineffective" for the following categories: Pain suppression (PS), speed of pain relief (SPR), duration of pain relief (DPR), general effectiveness (GE). Participants judged the treatment as "extremely useful, useful, not useful & could not be assessed" for overall evaluation (OE).
Time Frame: Baseline up to 8 hours post-administration of study treatment
Population: as for outcome 9
Measure: Number; unit: Percentage of participants
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Number analyzed (Participants) | 107 | 46 | 113
Percentage of participants
  PS:very effective (n=107, 46, 113) | 19.4 | 8.2 | 9.6
  PS:effective (n=107, 46, 113) | 2.8 | 0 | 0
  PS:somewhat effective (n=107, 46, 113) | 63.9 | 42.9 | 67.5
  PS:ineffective (n=107, 46, 113) | 13.9 | 49.0 | 22.8
  SPR:very effective (n=107, 46, 113) | 56.9 | 21.6 | 44.8
  SPR:effective (n=107, 46, 113) | 26.6 | 21.6 | 28.4
  SPR:somewhat effective (n=107, 46, 113) | 7.3 | 15.7 | 10.3
  SPR:ineffective (n=107, 46, 113) | 9.2 | 41.2 | 16.4
  DPR:very effective (n=41, 14, 53) | 39.0 | 28.6 | 24.5
  DPR:effective (n=41, 14, 53) | 26.8 | 35.7 | 28.3
  DPR:somewhat effective (n=41, 14, 53) | 17.1 | 7.1 | 20.8
  DPR:ineffective (n=41, 14, 53) | 17.1 | 28.6 | 26.4
  GE:very effective (n=107, 46, 113) | 2.8 | 0 | 0
  GE:effective (n=107, 46, 113) | 33.9 | 13.7 | 23.3
  GE:somewhat effective (n=107, 46, 113) | 46.8 | 31.4 | 53.4
  GE:ineffective (n=107, 46, 113) | 16.5 | 54.9 | 23.3
  OE:Extremely useful (n=107, 46, 113) | 0.9 | 0 | 0
  OE:useful (n=107, 46, 113) | 11.9 | 3.9 | 17.2
  OE:not useful (n=107, 46, 113) | 87.2 | 96.1 | 82.8
  OE:could not be assessed (n=107, 46, 113) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to Day 8
Description: An adverse event is any untoward medical occurrence in a clinical study participant administered with study treatment. It can be any unfavorable and unintended sign/abnormal finding, symptom, or disease temporally associated with the use of a medicinal (investigational) product, whether or not related to the medicinal (investigational) product.
Arm/Group | Tramadol Hydrochloride Plus Acetaminophen and Placebo | Tramadol Hydrochloride and Placebo | Acetaminophen and Placebo
Serious Adverse Events (participants affected / at risk) | 0/132 | 0/66 | 1/130
Other Adverse Events (participants affected / at risk) | 82/132 | 40/66 | 52/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride Plus Acetaminophen and Placebo (N=132) | Tramadol Hydrochloride and Placebo (N=66) | Acetaminophen and Placebo (N=130)
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tramadol Hydrochloride Plus Acetaminophen and Placebo (N=132) | Tramadol Hydrochloride and Placebo (N=66) | Acetaminophen and Placebo (N=130)
Alveolar osteitis (Infections and infestations) | 6 | 1 | 10
Post procedural infection (Infections and infestations) | 0 | 0 | 3
Nasopharyngitis (Infections and infestations) | 2 | 0 | 0
Urethritis (Infections and infestations) | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Somnolence (Nervous system disorders) | 39 | 15 | 14
Dizziness (Nervous system disorders) | 12 | 5 | 0
Headache (Nervous system disorders) | 7 | 5 | 4
Dizziness postural (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 0 | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 2 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Ear discomfort (Ear and labyrinth disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 20 | 10 | 4
Vomiting (Gastrointestinal disorders) | 10 | 2 | 1
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 4
Stomach discomfort (Gastrointestinal disorders) | 4 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 1 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0
Periodontitis (Gastrointestinal disorders) | 1 | 0 | 0
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 1
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Gastric disorder (Gastrointestinal disorders) | 0 | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Swelling face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Feeling abnormal (General disorders) | 4 | 5 | 1
Pyrexia (General disorders) | 4 | 1 | 1
Malaise (General disorders) | 2 | 0 | 0
Asthenia (General disorders) | 1 | 0 | 0
Chills (General disorders) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 12 | 6 | 11
White blood cell count increased (Investigations) | 2 | 2 | 2
Blood triglycerides increased (Investigations) | 0 | 1 | 1
Blood urea increased (Investigations) | 1 | 1 | 0
Protein urine present (Investigations) | 1 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1
Blood creatinine increased (Investigations) | 0 | 1 | 0
Blood potassium decreased (Investigations) | 1 | 0 | 0
Blood pressure increased (Investigations) | 0 | 1 | 0
Blood uric acid increased (Investigations) | 0 | 1 | 0
Glucose urine present (Investigations) | 0 | 1 | 0
Blood urine present (Investigations) | 0 | 0 | 1
Liver function test abnormal (Investigations) | 1 | 0 | 0
Mouth injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the Principal Investigator is that the Sponsor can review results communications prior to public release.